CLINICAL TRIAL: NCT04777279
Title: Physical Exercise and Nutrition Supplement on Improving Frailty, Depressive Symptoms, and Quality of Life in Community-dwelling Older Population
Brief Title: Physical Exercise, Nutrition Supplement and Frailty of Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, associate professor, Taipei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202010046
Record Dates: First submitted 2021-01-26; First posted 2021-03-02 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Physical Exercise; Nutrition Poor; Elderly
MeSH Terms: conditions — Sarcopenia; Motor Activity; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Individual physical exercise group (Experimental): a 12-weeks physical exercise program (60 minutes/ three times weekly)
  Interventions: Behavioral: individual physical exercise group
- Individual Branched-Chain Amino Acids supplements group (Experimental): a 12-weeks Branched-Chain Amino Acids supplements (5 g Branched-Chain Amino Acids every day)
  Interventions: Dietary Supplement: individual Branched-Chain Amino Acids supplements group
- Combination of physical exercise and Branched-Chain Amino Acids supplements group (Experimental): a 12-weeks physical exercise program (60 minutes/ three times weekly) and a 12-weeks Branched-Chain Amino Acids supplements (5 g Branched-Chain Amino Acids every day)
  Interventions: Other: combination of physical exercise and nutrition supplements group
- Control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: individual physical exercise group — The participants in physical exercise group will receiving individual physical exercise lead by physiological therapist for 60 minutes/ three times weekly for 12 weeks.
  Arms: Individual physical exercise group
Dietary Supplement: individual Branched-Chain Amino Acids supplements group — The participants in nutrition supplements group will receiving Branched-Chain Amino Acids 5 g Branched-Chain Amino Acids every day for 12 weeks.
  Arms: Individual Branched-Chain Amino Acids supplements group
Other: combination of physical exercise and nutrition supplements group — The participants in physical exercise group will receiving physical exercise lead by physiological therapist for 60 minutes/ three times weekly for 12 weeks and 5 g Branched-Chain Amino Acids every day for 12 weeks.
  Arms: Combination of physical exercise and Branched-Chain Amino Acids supplements group

SUMMARY:
This study is aimed to explore the effect of physical exercise and nutrition supplement on improving frailty, depressive symptoms, and quality of life in community-dwelling older population.

DETAILED DESCRIPTION:
Objective: This study is aimed to explore the effect of physical exercise and nutrition supplement on improving frailty, depressive symptoms, and quality of life in community-dwelling older population.

Methods: We conduct a quasi-experimental study to measure frailty, depressive symptoms, and quality of life before and after intervention. A total of 120 community-living older adults with frailty identified by Fried's phenotype method are assigned to four groups: physical exercise group, nutrition supplements group, physical exercise and nutrition supplements group, and control group. Each participants in the assigned group will receive 12 weeks intervention. Measurements include frailty (Fried's phenotype method), depressive symptoms (Geriatric Depression Scale-15, GDS-15), and quality of life (WHOQOL-BREF). Data analyses include describe statistics, Chi-square test, and Analysis of Variance. A Generalized estimating equations (GEE) will be used to examine the effect of physical exercise and nutrition supplement on improving frailty, depressive symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged more than 60 years;
* pre-frail stage: must have one item as frailty identified using the Fried's phenotype method;
* normal cognition: AD8 score less than 2 points;
* can communicate with Mandarin or Taiwanese.

Exclusion Criteria:

* incapable of walk independent or using assistive devices (e.g., crutches);
* a condition of having an acute disease, hemodialysis, or unable to engage in physical activity;
* have history of unstable heart disease such as coronary heart disease, heart failure and hypertension without regular medication;
* have regular physical activity (≥150 minutes weekly) such as aerobic dance, swimming, Tai Chi.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
frailty score | frailty score at baseline
  Frailty will examined using Fried's phenotype method and higher score indicates more frailty
frailty score | through study completion, an average of 12 weeks
  Frailty will examined using Fried's phenotype method and higher score indicates more frailty

SECONDARY OUTCOMES:
Depressive symptoms score | Depressive symptoms at baseline
  Depression will measured using Geriatric Depression Scale-15 (GDS-15) and and higher score indicates more depression
Depressive symptoms score | through study completion, an average of 12 weeks
  Depression will measured using Geriatric Depression Scale-15.
Quality of Life score | Quality of Life at baseline
  Quality of Life will examined using World Health Organization Quality of Life scale and higher score indicate better quality of life
Quality of Life score | through study completion, an average of 12 weeks
  Quality of Life will examined using World Health Organization Quality of Life scale and higher score indicate better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen LF, Chang HC, Cai ZC, Chen YJ, Hsu WL, Chuang YH, Lee SC, Huang HC. Community-based exercise and nutritional interventions to improve frailty syndrome among older adults: A quasi-experimental study. Geriatr Nurs. 2023 May-Jun;51:222-231. doi: 10.1016/j.gerinurse.2023.03.016. Epub 2023 Apr 3. PMID 37018848